CLINICAL TRIAL: NCT03632863
Title: Randomized Controlled Trial of an Electronic Patient Decision Aid (PDA) for Antidepressant Medication Use in Pregnancy
Brief Title: PDA for Antidepressant Use in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Simone Vigod, Psychiatrist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-0069-B
Record Dates: First submitted 2018-07-31; First posted 2018-08-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Depression
Keywords: Pregnancy; Depression; Antidepressant Use; Decision Aid
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Patient Decision Aid (Experimental): Participants login to a website where they access the interactive PDA as well as access standard published information and resources.
  Interventions: Behavioral: Electronic Patient Decision Aid; Behavioral: Standard Resource Sheet
- Standard Resource Sheet (Sham Comparator): Participants login to a website where they access standard published information and resources.
  Interventions: Behavioral: Standard Resource Sheet

INTERVENTIONS:
Behavioral: Electronic Patient Decision Aid — The electronic PDA is an interactive website with 3 main sections:
  1. Review of depression treatment options (non-pharmacological and pharmacological) along with their respective risks and benefits.
  2. Interactive "values clarification" exercises to help women determine which risks and benefits are most important to them.
  3. Exercises to help women consider how partners, family, providers and the social context impacts decision-making.
  A summary of how a woman feels about each option along with risks and benefits is generated which can be provided to treating clinicians for use in follow-up.
  A printable pdf with standard published information and resources is also included.
  Arms: Electronic Patient Decision Aid
Behavioral: Standard Resource Sheet — A control group aims to isolate the PDA's effects from time and clinical care. Controls login to the study website and receive the same printable pdf as in the PDA so that they can access standard publicly available information/resources, even if they will not receive the PDA.

SUMMARY:
Depression in pregnancy is common, affecting up to 10% of women and represents serious risk to mother and infant. Unfortunately, antidepressant medication, a first-line treatment for depression in pregnancy, also comes with risks, making this a complex decision. Clinical care appears to be insufficient for ensuring that women make decisions that are consistent with their own values and with which they feel satisfied. Patient decision support tools can address such barriers. We have created and piloted with positive results an online patient decision aid (PDA) that has the potential to improve the decision-making process for women regarding antidepressant use in pregnancy in conjunction with clinical care. The overall objective of this study is to conduct a Randomized Controlled Trial (RCT) to assess the efficacy of our PDA for antidepressant use in pregnancy.

DETAILED DESCRIPTION:
A parallel group randomized controlled trial (RCT) will be conducted. Eligible and consenting women with depression will be randomized in a 1:1 ratio to either online PDA or a control condition comprising an online set of publicly available standard resources. The study will be stratified by preconception vs. pregnant, and by province.

The study is based at Women's College Hospital (Toronto) but participants will be recruited from across Canada, as the online intervention does not require any in-person study visits. Participants will be recruited via social media (ex. Facebook, Twitter, mommy/baby blogs) and by provider referrals.

Participants will be given a series of online questionnaires with various measures collected at baseline, 4 weeks post-randomization, in each trimester of pregnancy, and at 1, 3, 6 and 12 months postpartum. Participants who are planning pregnancy will enter the longer-term (pregnancy and postpartum) follow-up phase once they become pregnant; those who do not conceive by one year post-randomization will be sent a final set of questionnaires and exit the study. A process evaluation will also be conducted to gain insights around trial conduct, and perspectives on potential for (or barriers to) scale-up. This, along with the planned economic evaluation, will inform clinical and policy decisions around adopting the PDA into real-world practice.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 18 years old; and
2. Diagnosed with major depressive disorder (current or in remission); and
3. Planning conception in the next 12 months or < 30 weeks gestational age; and
4. Deciding whether to start or continue a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) in pregnancy; and
5. Have moderate-to-high decisional conflict regarding the decision to start or continue an SSRI/SNRI in pregnancy; and
6. Live in Canada

Exclusion Criteria:

1. Have had alcohol or substance use disorder in prior 12 months; or
2. Have active suicide ideation or psychosis; or
3. Have past/current major obstetrical or fetal complications; or
4. Are unable to complete relevant study procedures online; or
5. Are unable to complete study procedures in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Postpartum depression as diagnosed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (SCID-I) | 3 months postpartum
  The depression module will be used to indicate presence of postpartum depression.

SECONDARY OUTCOMES:
Postpartum depression as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-I) | 12 months postpartum
  The depression module will be used to indicate presence of postpartum depression.
Maternal knowledge of depression, postpartum depression and antidepressant use during pregnancy | baseline and 4 weeks
  True/false knowledge questionnaire.
Decisional conflict as measured by the Decisional Conflict Scale (DCS) | throughout pregnancy (up to 9 months)
  DCS consists of 16 items each rated 1-5 where scores ≥ 25 represent delayed and ineffective decisions.
Maternal depression as measured by the Edinburgh Postnatal Depression Scale (EPDS) | throughout pregnancy and up to 1 year postpartum (up to 21 months)
  EPDS is a 10-item self-report scale. Each item is scored 0-3 with scores >12 being predictive of a diagnosis of depression.
Maternal anxiety as measured by the Spielberger State-Trait Anxiety Inventory (STAI) | throughout pregnancy and up to 1 year postpartum (up to 21 months)
  STAI is a 40-item self-report scale with good discriminate validity in perinatal populations. Each item is scored 1-4 with scores >48 being predictive of an anxiety disorder diagnosis.
Maternal quality of life as measured by the 12-item Short Form (SF-12) Health Survey | throughout pregnancy and up to 1 year postpartum (up to 21 months)
  SF-12 is a 12-item survey used to estimate the quality-adjusted life year (QALY) which incorporates both length of life and quality of life into a single measure. The measure includes a physical component summary and a mental component summary score. It is scored 0-100 with higher scores indicating better physical and mental health.
Study website metrics to inform if patterns of PDA use are predictive of clinical outcomes | throughout pregnancy (up to 9 months)
  Data generated by the website to inform how participants interact with the PDA: 1) proportion of participants who login to the PDA; 2) timing from enrollment to first login; 3) total number of PDA logins; 4) number of logins between each study time point; 5) proportion of participants who completed the PDA; 6) timing of enrollment to first completion of PDA; 7) number of logins required prior to first completion of PDA; 8) total number of PDA completions; 9) number of PDA completions between each study time point; 10) mean (SD) number of pages viewed per login; 11) whether or not each page was viewed; 12) whether or not each page was viewed between study time points; 13) whether or not each interactive tag was interacted with; 14) whether each interactive tag was interacted with between study time points
Health service utilization | throughout pregnancy and up to 1 year postpartum (up to 21 months)
  1) direct medical costs; 2) indirect medical costs; 3) productivity loss due to patient and family work absence
Pregnancy complications and neonatal outcomes | 1 month postpartum
  Self-reported pregnancy complications and neonatal infant characteristics
Infant Outcomes as measured by the Infant Characteristics Questionnaire (ICQ) | 3-12 months after birth
  ICQ is a 27-item questionnaire with each item scored 1-7. Higher scores indicate higher parental perceptions of difficult infant temperament.
Child Development as measured by the Ages and Stages Questionnaire (ASQ-3) | 3-12 months after birth
  ASQ-3 is a 30-item instrument that screens for child development from 1 to 60 months. Items are scored as 0, 5 or 10 points. Higher scores indicate that the child is doing well.
Parenting stress measured by the Parenting Stress Index (PSI) short form | 1 month postpartum to 1 year postpartum
  The PSI-SF is a 36-item measure consisting of 3 subscales (parental distress, dysfunction in parent-child relations, difficult child). Each item is scored 1-5 with higher scores indicating higher levels of parenting stress. PSI reports subscales separately and also reports a total measure.
Partner relationship outcomes measured by the Dyadic Adjustment Scale (DAS) | throughout pregnancy and up to 1 year postpartum (up to 21 months)
  DAS is a self-report measure of relationship adjustment. An abbreviated version of this scale consisting of only the dyadic consensus subscale will be used. Each item is scored 0-5 with higher scores indicating a higher level of agreement amongst couples.
Bipolar disorder as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-I) | 3 months and 12 months postpartum
  The bipolar disorders module will be used.
Schizophrenia and other psychotic disorders as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-I) | 3 months and 12 months postpartum
  The schizophrenia and other psychotic disorders module will be used.
Anxiety disorders as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-I) | 3 months and 12 months postpartum
  The anxiety disorders module will be used.
Obsessive-compulsive and related disorders as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-I) | 3 months and 12 months postpartum
  The obsessive-compulsive and related disorders module will be used.
Feeding and eating disorders as diagnosed by the Structured Clinical Interview for DSM-5 (SCID-I) | 3 months and 12 months postpartum
  The feeding and eating disorders module will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Vigod, MD, MSc, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No